CLINICAL TRIAL: NCT03203954
Title: Neural Substrates of Reinforcement Learning and Its Training in Major Depression
Brief Title: Testing the Neuroscience of Guided Learning in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Pearl Chiu, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MDDLEARNING; R01MH106756 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Training (Active Comparator): Guided learning, standard learning: Repeat administration of standard behavioral learning task
  Interventions: Behavioral: Standard Learning
- Instructed Statistics (Experimental): Guided learning, instructed statistics: Repeat administration of behavioral learning task with instructions about task statistics
  Interventions: Behavioral: Guided Learning: Instructed statistics
- Not Instructed Statistics (Experimental): Guided learning, changing statistics: Repeat administration of behavioral learning task with changing task statistics
  Interventions: Behavioral: Guided Learning: Changing statistics

INTERVENTIONS:
Behavioral: Standard Learning — Participants will complete repeat sessions of a computer-based learning task, and task performance and symptoms will be assessed.
  Arms: No Training
Behavioral: Guided Learning: Instructed statistics — Participants will complete repeat sessions of a computer-based learning task, and task performance and symptoms will be assessed.
  Arms: Instructed Statistics
Behavioral: Guided Learning: Changing statistics — Participants will complete repeat sessions of a computer-based learning task, and task performance and symptoms will be assessed.
  Arms: Not Instructed Statistics

SUMMARY:
Major depression is a prevalent and impairing illness. To better understand the basic science and treatment of depression, the investigators study the behavioral and brain processes associated with learning in depression and how potential disruptions in learning may be repaired. Understanding different methods that change learning may lead to novel treatments that contribute to recovery in people with depression.

DETAILED DESCRIPTION:
Major depressive disorder ranks among the most significant causes of mortality and disability in the world. Recent data from the investigators and others highlight that impairments in reward and loss learning are central to depression, have distinct neural substrates, and improve with successful treatment. Together, these findings suggest an urgent need to delineate the relationships among neural and behavioral learning impairments and depression. Equally important, these insights suggest new targets for treatment such that manipulating the neural and behavioral substrates of learning may facilitate symptom change in depression.

To address these issues, the investigators use functional neuroimaging and a computational psychiatry framework to i) systematically characterize the neural and behavioral substrates that attend reward- and loss- learning in depression and ii) assess the degree to which learning in depression responds to two behavioral methods that target learning in different ways. The investigators test the broad hypotheses that i) that depression may be characterized by distinct neural and behavioral disruptions of learning, and ii) these disruptions and associated symptoms may be ameliorated through different methods of guiding learning. Recent advances in computational psychiatry provide a mechanism-based framework within which to understand the nature and trajectory of potential learning impairments in depression and suggest new ways that disrupted learning and associated symptoms may be improved in depression

ELIGIBILITY:
Inclusion Criteria:

* males and females of all ethnicities
* meet diagnostic criteria for major depression or non-depressed control (assessed by study staff)
* ages 18-55
* fluent in English
* able to see computer display clearly
* able to provide informed consent
* able to follow verbal or written instructions
* for participants who are referred by a clinician, a letter from that clinician indicating that participation in the study does not constitute an elevated medical or behavioral risk to the participant will be requested.

Exclusion Criteria:

* current pregnancy or menopause
* claustrophobia
* MRI contraindications
* psychotic or bipolar disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Task performance | approximately 6 weeks (pre- post- learning task changes and interim time points)
  behavioral measures of learning task performance including accuracy, learning rate

SECONDARY OUTCOMES:
Neuroimaging measures | approximately 6 weeks (pre- post- learning task changes and interim time points)
  functional MRI during learning task performance
Symptoms | approximately 6 weeks (pre- post- learning task changes and interim time points)
  self-report questionnaires and clinician-obtained symptom measures

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Tech Carilion Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
following study completion, de-identified data will be made available to approved researchers and may be requested from the principal investigator